CLINICAL TRIAL: NCT06606977
Title: The Impact of 8-week Re-training Following a 14-week Period of Detraining on Greco-Roman Wrestlers
Brief Title: The Impact of Re-training Following Detraining on Greco-Roman Wrestlers
Status: Completed | Type: Observational
Sponsor: Tuba Melekoğlu (Other)
Responsible Party: Sponsor-Investigator, Tuba Melekoğlu, Assoc. Prof., Akdeniz University
Organization: Akdeniz University (Other)
Other Study IDs: TYL-2021-5677
Record Dates: First submitted 2024-09-16; First posted 2024-09-23 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Heart Rate Variability; Body Fat; Wrestling; Fitness Testing
Keywords: Wrestling; training; detraining; heart rate variability

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 16 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Elite Greco-Roman Wrestlers: Elite senior wrestlers in the Greco-Roman style participated in the study. These wrestlers had not participated in field training for a minimum of 14 weeks due to the Covid-19 epidemic, and this study focuses on their performance and autonomous system response after resuming field training.
  Interventions: Other: Training

INTERVENTIONS:
Other: Training — During the detraining period, the athletes did not follow any external (personal) trainer-supported training program and their diet was not altered. Athletes have reported that they have stayed at home as a necessity of the Covid-19 pandemic process, and have done simple home exercises, walking and jogging exercises in a limited way during this time.
  The training period included the standard wrestling trainings, which were determined by the national team coaches and realized at different intensities, during the 8 weeks when the training started. Following the period of detraining the level of training intensity was progressively increased throughout the initial 5 weeks. In the 6th and 7th week, training intensity peaked . In the 8th week prior to the competition, the training intensity was reduced in order to prepare and recover for the following competition. After the training period, the wrestlers participated in an international competition.
  Other Names: Wrestling training and conditioning; Detraining

SUMMARY:
The aim of this study is to analyse the alterations in the physical, physiological, and performance characteristics of the elite Greco-Roman wrestlers who experienced a prolonged period of detraining (14 weeks) as a result of the Covid-19 pandemic. Elite Greco-Roman wrestlers volunteered for the research. Heart rate variability values were measured during the detraining period and for 8 weeks of subsequent training, and then interpreted for training periods with different workloads. Body fat percentage measured during detraining and every 2-week interval during the training period. To determine the fitness status of wrestlers, the Specific Wrestling Fitness test was used before and following the 8-week training period.

DETAILED DESCRIPTION:
Elite athletes train continuously and at high intensity in a planned and regular basis in order to achieve success in the international competitions in line with the necessity of the competitive conditions, to maintain the success achieved and to preserve it for a long time. As a result of these high-intensity training, the physiological adaptations of elite athletes are different when compared to sedentary individuals and other athletes. For this reason, athletes who want to show high performance take care to maintain these adaptations as well as develop them. In addition, it is necessary to provide training stimuli at a regular and sufficient level in order to maintain or develop these adaptations Excessive training stimulus can lead to overtraining, while inadequate or complete cessation of training can result in a loss of performance known as detraining.

High-level competitive athletes who do not want to experience this loss of performance avoid taking a long break from training by limiting the detraining period. However, in some cases (injury, chronic injury, pregnancy in female athletes, etc.) athletes are forced to enter a detraining period. In these cases of partial or complete cessation of training, it is predicted that the organism's response time to exercise is prolonged. In case of interruption of training for up to 4 weeks, decreases can be seen in general endurance and muscular endurance performance without significant changes in muscle strength, while losses in muscle strength are seen in addition to muscle endurance in periods exceeding four weeks 3. Research indicates that after a detraining period, there is a tendency for skinfold thickness, body fat mass, and percentage to increase, and for fat-free mass and athletic performance to decrease. On the other hand, literature says that athletes can regain their muscle strength in a short time after short-term (3 weeks) detraining. Yasuda et al. reported that as a result of the strength training practices applied with the blow flow restriction method after 3 weeks of detraining to individuals who had previously done strength training, muscle strength gains were rapidly achieved.

In addition to physical losses such as strength and endurance in the organism, the autonomic nervous system (ANS), which is an indicator of general health and an important reflector of optimal sportive performance in athletes, and heart rate variability scores, which are frequently used to determine ANS, may also show negative deterioration in the event of cessation of exercise. A prolonged period of detraining can cause significant deterioration in heart rate variability values and is often associated with a decreased athletic performance.

In early 2020, a worldwide outbreak of coronavirus disease has occurred, which is considered a global emergency. Preventive strategies aimed at minimizing the risk of infection include the utilization of social gatherings. The impact on elite sport has been significant, with ongoing championships halted and major international events postponed. Moreover, the majority of elite athletes are forced to participate in isolated and usually unsupervised training sessions within the boundaries of their own homes. Following the lockdown, it was recommended that trainings be carefully planned and that performance and health parameters be closely watched to ensure a safe return to the competitions. This approach helped prevent injuries and allowed athletes to gradually regain their physical condition.

Although there are some studies on the effects of long-term inactivity on physical and physiological adaptations and sports performance parameters in elite athletes, there are not enough studies on elite wrestlers that examine the effects of such prolonged inactivity (14 weeks) on their physical and physiological recovery levels recovery and the present knowledge of the period required for elite-level wrestlers to attain optimal performance levels in getting ready for potential competitions remains inadequate.

The purpose of this study was to examine the changes in the physical and physiological conditions of elite wrestlers on the Turkish National Wrestling Team who were exposed to physical inactivity for 14 weeks after the Covid-19 pandemic lockdown, followed by an 8-week training and competition period.

ELIGIBILITY:
Inclusion Criteria:

* Being 19 years or older
* An elite athlete who had international competition experience
* Not taking any medication that may affect cardiac capacity
* Absence of a disease that may affect the cardiac or autonomic nervous system.

Exclusion Criteria:

* Desire to leave the study
* Failure to participate measurements for concurrent 5 days
* Injury or long-term illness during training period.

Min Age: 19 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study included 20 male volunteer wrestlers who were members of the national wrestling team and had been training for 10 years. The wrestlers in the research group consisted of elite level athletes. Two of them had European and World championship medals and 7 of them had other medals in the year before the untrained period. In the year after the untrained period, one of these athletes won world silver medal and the following year gold medal. In addition, 6 of the athletes won medals at the European and World Championships.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2021-08-09 (Actual); Primary Completion 2023-04-19 (Actual); Study Completion 2023-04-19 (Actual)

PRIMARY OUTCOMES:
Heart Rate Variablity | From enrollment to the end of treatment at 16 weeks
  The measurements included evaluating the intervals between the QRS complexes, executing statistical analyses such as SDNN and RMSSD, and performing frequency-domain analyses including LF, HF, and LF/HF

SECONDARY OUTCOMES:
Body Fat Percentage | From enrollment to the end of treatment at 8 weeks
  Body fat percentage was measured with bioelectrical impedance and skinfold caliper
Specific Wrestling Fitness Test Performance | From enrollment to the end of treatment at 8 weeks
  The SWFT includes throwing maximum wrestling dummy against time. Since wrestling is a sport based on weight categories, participants should use a wrestling dummy suitable for their own weight (wrestlers up to 74.9 kg body weight a 22 kg dummy, wrestlers from 75.0 to 89.9 kg a 27 kg dummy and for wrestlers over 90 kg a 32 kg dummy). The participant was performed three sets of dummy throws lasting 30 seconds each, with a 20-second interval of rest between each set. Following the start signal, the participants were attempted to throw the wrestling dummy repeatedly within the given 30-second timeframe, using maximum effort. The primary objective of the participant was to execute as many throws possible in all three phases of the tests, with the cumulative number of throws executed providing as the final test outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Tuba Melekoglu, Phd, Principal Investigator — Akdeniz University
Locations (1):
- Akdeniz University Faculty of Sport Sciences, Antalya, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
all IPD collected throughout the trial will be shared
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Will be available 10 September 2024
Access Criteria: The datasets generated during the current study will be available upon request from corresponder author Tuba Melekoğlu

REFERENCES:
- [Background] Alvurdu S, Baykal C, Akyildiz Z, Senel O, Silva AF, Conte D, Clemente FM. Impact of Prolonged Absence of Organized Training on Body Composition, Neuromuscular Performance, and Aerobic Capacity: A Study in Youth Male Soccer Players Exposed to COVID-19 Lockdown. Int J Environ Res Public Health. 2022 Jan 20;19(3):1148. doi: 10.3390/ijerph19031148. PMID 35162174